CLINICAL TRIAL: NCT03016390
Title: Electromagnetic Interference and Automobile Remote Keyless Entry in Cardiovascular Implantable Electronic Device (CIED) Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chiang Mai University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Narawudt Prasertwitayakij, lecturer, Chiang Mai University
Other Study IDs: MED-2559-03815
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Electromagnetic Interference in Cardiovascular Implantable Electronic Device
Keywords: Cardiac Implantable Electronic Device; Pacemaker; Automatic Implantable Cardioverter-Defibrillator (AICD); Electromagnetic interference (EMI); Keyless access system; Keyless entry system

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
Cardiovascular Implantable Electronic device (CIED) is a evolution therapy and number of patients with it are growing rapidly. Electromagnetic interference causing device malfunction is not uncommon, Radiofrequency Identification system is among its plausible source. Patients with CIEDs are at risk of exposure to this novel product in their daily living especially automobile keyless access system. Only informal studies have been conducted and not be published. Formal and systemic evaluation and tests are crucial.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years old
2. Able to give informed consent
3. Implanted with functioning pacemakers or AICD more than 3 months
4. Adequate and stable all device parameters
5. Able to operate self triggering event recorders (at least 30 seconds)

Exclusion Criteria:

1. Patient with single chamber (Atrial) pacemaker (AAI or AAIR)
2. Presence of unstable hemodynamic or conditions
3. Presence of sustained or ongoing arrhythmia, besides atrial fibrillation/atrial flutter in single (ventricle) chamber device or Atrio-ventricular block
4. Documented of over-sensing episodes under regular sensitivity threshold (0.25 mV or more in the atrial channel and 0.75 mV or more in the ventricular channel, for permanent pacemaker device, and manufacture default setting in Automatic Implantable Cardioverter-Defibrillator, AICD)
5. Lack of noise oversensing detection/trigger and Electrogram (EGM) storage capability
6. Lack of tachyarrhythmia detection and episode storage capability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients participated at our Cardiac Rhythm Device Management (CRDM) clinic at Maharaj Nakorn Chiang Mai hospital, Faculty of medicine, Chiang Mai University will be invited. And at least 100 consecutive patients to be equally enrolled in both pacemakers(including single chamber, dual chamber and Cardiac Resynchronization Therapy pacemaker-CRTP) and Automatic Implantable Cardioverter-Defibrillator (AICD) (including single chamber, dual chamber and Bi-ventricular AICD or CRTD)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of any Electromagnetic interference | Immediately after completion of the protocol test

SECONDARY OUTCOMES:
Incidence of pacing inhibition in ventricular channel | Immediately after completion of the protocol test
Incidence of noise reversion | Immediately after completion of the protocol test
Incidence of ventricular tachycardia/fibrillation detection | Immediately after completion of the protocol test

CONTACTS AND LOCATIONS:
Overall Officials: Arintaya Phrommintikul, MD, Study Chair — Faculty of Medicine, Chiang Mai University

REFERENCES:
- [Derived] Prasertwitayakij N, Komolmis T, Gunaparn S, Pisespongsa C, Phrommintikul A, Wongcharoen W, Nantsupawat T. Electromagnetic interference from automobile passive keyless entry in cardiovascular implantable electronic devices. Expert Rev Med Devices. 2023 Jul-Dec;20(11):973-977. doi: 10.1080/17434440.2023.2255126. Epub 2023 Sep 5. PMID 37668539